CLINICAL TRIAL: NCT04022798
Title: Randomized Controlled Trial of Effectiveness of Neural Mobilization in the Management of Chronic Low Back Pain With Radiculopathy.
Brief Title: Management of LBP With Radiculopathy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tabuk (Other)
Responsible Party: Principal Investigator, Salem F Alatawi, Clinical Professor, University of Tabuk
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTabuk
Record Dates: First submitted 2019-07-08; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Low Back Pain
Keywords: Low back pain; Neural mobilization; lumbar stabilization exercise; Radial extracorporeal shock wave therapy
MeSH Terms: conditions — Low Back Pain | interventions — Exercise; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Experimental group: Group A (NM, LSE and rESWT) and Control group: Group B (LSE and rESWT).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Neural mobilization (NM), lumbar stabilization exercise (LSE) and Radial Extracorporeal Shock Wave Therapy (rESWT)
  Interventions: Other: Exercise, manual therapy
- Control group (Active Comparator): lumbar stabilization exercise (LSE) and Radial Extracorporeal Shock Wave Therapy (rESWT)
  Interventions: Other: Exercise, manual therapy

INTERVENTIONS:
Other: Exercise, manual therapy — Participants were randomly assigned into treatment (n=15) or control group (n=15). Participants in each group received 12 treatment sessions of 45 minutes each, 2 days a week for 6 consecutive weeks.
  For each group, a menu of a lumbar stabilization program was designed. This program included 8 levels of exercise ( single leg knee to chest stretch, double leg knee to chest, supine piriformis stretch, supine hamstring stretch, lower trunk rotation stretch, lumbar rotation stretch, pelvic tilt, pelivic tilt with alternative legs). Exercises were tailored for each individual ability and, if possible, progressed at each session which would last approximately 30 minutes. Each single exercise was repeated many times based on the patient's clinical condition. All sessions were provided by physiotherapists.

SUMMARY:
This study is to determine the effectiveness of Neural mobilization(NM) technique compared with lumbar stabilization exercise (LSE) and Radial Extracorporeal Shock Wave Therapy (rESWT) in the physical therapy management of chronic low back pain (CLBP) with radiculopathy. Subjects will be randomly assigned into two groups. Group A (NM, LSE and rESWT) and Group B (LSE and rESWT).

DETAILED DESCRIPTION:
Randomized clinical control trail will be conducted in the North West area of Saudi Arabia.

Patients diagnosed to have CLBP with radiculopathy at three different hospitals in Saudi Arabia will be recruited for this study.

Participants will be randomly assigned into treatment or control group. Before starting of the study, the author will designe the treatment and control group treatment program and instructed the treating physiotherapists in their implementation. An ethical approval was approved by the ethics committee of the University of Tabuk- Saudi Arabia. Participants in each group will receive 12 treatment sessions of 45 minutes each, 2 days a week for 6 consecutive weeks.

For each group, a menu of a lumbar stabilization program was designed. This program included 8 levels of exercise ( single leg knee to chest stretch, double leg knee to chest, supine piriformis stretch, supine hamstring stretch, lower trunk rotation stretch, lumbar rotation stretch, pelvic tilt, pelivic tilt with alternative legs). Exercises were tailored for each individual ability and, if possible, progressed at each session which would last approximately 30 minutes. Each single exercise was repeated many times based on the patient's clinical condition. All sessions were provided by physiotherapists. After finishing of session of lumbar stabilization program, a shock wave therapy was applied for each participant in a prone position over the region of low back pain (Figure 2 ).

Only participants in the treatment group were receive neural mobilization technique. This includes the following: sciatic neural mobilization technique (Figure 3), slump neural mobilization technique (Figure 4) and self neural mobilization (Figure 5 ).

OUTCOME MEASUREMENT TOOLS:

There were three outcome measures as following: pain, disability and lumbar spine range of motion. Subjected were tested three times as following: at the baseline (0 week), at the mid of treatment (3 weeks) and finally at the end of treatment (6 weeks).

* Pain Pain was assessed by using NPRS, where 0 represented no pain and 10 represented the worst pain possible, to indicate the intensity of pain in the lower back (Jensen et al., 1994). Disability Disability was measured by using the Modified Oswestry Disability Questionnaire (MODQ) which is a self-rating questionnaire used to evaluate functional physical disability (Rajfur, et al., 2017).
* Lumbar flexion range of motion Lumbar flexion range of motion was measured by using modified Schober method (Philadelphia Panel Members, 2001).

DATA ANALYSIS:

A simple descriptive statistical analysis was adopted to describe the patient specific demographic characteristics with respect to outcomes parameters. Within group and between groups comparison was analyzed using ANOVA and Scheffes' post-hoc tests by using SPSS 20.0.

Work Plan:

Roles and responsibilities :

1. Principal Investigator-is responsible for the following:

1. The management and integrity of the research design 2. Approval from ethical board committee or its equivalent 3. Preparation and conduct of the study 4. Reporting of the research project 5. Managing, monitoring and ensuring the integrity of any collaborative relationships.

6. Directs and oversees compliance, financial, personnel, and other related aspects and resources of the research project 7. Coordination with department and central administration personnel to assure research in is conducted in accordance with regulations of the University and sponsoring agency policies and procedures.

8. Publication of the study, local and international. Work Flow

1. The principal investigator will be responsible in check points, meetings, and coordination with the research team, regular meeting will be set on thursday every after two weeks and when necessary.
2. Co-investigator will be assigned as custodian to all data and investigations from the start of the study.
3. Co-investigator will be assigned to record all financial transaction according to the policies of sponsoring unit of the university.
4. Co-investigator will be responsible logistic and making sure all researched needed are adequate and available when needed.
5. A clear communication and coordination scheme will be established.
6. Co-investigator will be required to submit status accomplish report on regular basis determined by the team.

Utilization:

The outcomes of the research will be used to:

* NM techniques enhance patient outcomes in the management of CLBP with radiculopathy when added to standard care.
* NM technique applied by experienced physical therapists combined with LSE and ESWT in a brief clinical trial might better and earlier than LST and ESWT alone for decreasing pain, reducing back disability and improving function in patients with CLBP with radiculopathy symptoms.
* The findings are interesting and motivate further studies, including long-term follow-up of large groups, randomized studies and the comparison of this treatment model with other treatment models.
* A faster program with fewer hospital visits not only enables the patients to proceed with most of their daily activities but also decreases the costs of the treatment.
* A NM technique might also be an alternative to conventional physiotherapy in the treatment of the CLBP patients with radiculopathy symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Lower back pain should be Lower than 5 on the Visual Analogue Scale,
* > 18 years,
* Not taken physical therapy treatment in the past 6 months period,
* No previous surgery, such as structural anomalies, spinal cord compressions, severe instabilities, severe osteoporosis, acute infections, severe cardiovascular or metabolic diseases,
* A body mass index less than 30kg/m2.

Exclusion Criteria:

* Pain with a score above 5 on the Visual Analogue Scale (VAS),
* ≤ 18 years,
* Had physical therapy treatment in the past 6 months period,
* Had undergone previous surgery, such as structural anomalies, spinal cord compressions, severe instabilities, severe osteoporosis, acute infections, severe cardiovascular or metabolic diseases,
* pregnant
* A body mass index above 30kg/m2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain is being assessed using NPRS | baseline, 3 weeks and 6 weeks
  Pain was assessed by using NPRS, where 0 represented no pain and 10 represented the worst pain possible, to indicate the intensity of pain in the lower back (Jensen et al., 1994).
Change in Disability is being assessed using the Modified Oswestry Disability Questionnaire | baseline, 3 weeks and 6 weeks
  Disability was measured by using the Modified Oswestry Disability Questionnaire (MODQ) which is a self-rating questionnaire used to evaluate functional physical disability (Rajfur, et al., 2017).
Change in Lumbar flexion range of motion is being assessed using modified Schober method | baseline, 3 weeks and 6 weeks
  Lumbar flexion range of motion was measured by using modified Schober method (Philadelphia Panel Members, 2001).

CONTACTS AND LOCATIONS:
Overall Officials: Salem F Alatawi, PhD, Principal Investigator — University of Tabuk
Locations (1):
- Salem F Alatawi, Tabuk, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
After publication